CLINICAL TRIAL: NCT07033065
Title: In Hospital and Long Term Outcomes After Recurrent Ventricular Arrythmias
Brief Title: Recurrent Ventricular Arrythmias in ICU
Acronym: ElectStorm
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Principal Investigator, Batric POPOVIC, Professor, Central Hospital, Nancy, France
Other Study IDs: 2023PI147
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Ventricular Arrythmia; Cardiogenic Shock; Electrical Storm
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Electrical storm (ES) is a life-threatening syndrome defined by the recurrence of ventricular arrythmias.

ES is also represented by a wide spectrum of clinical situations ranging from recurrent monomorphic VT reduced by anti-tachycardia pacing (ATP) in relatively stable patients to recurrent VF in hemodynamically unstable patients.

Thus, the purpose of this study was to assess the incidence and predictors of long term mortality following hospitalization in the intensive care unit for ES, in a large retrospective multicentric study.

DETAILED DESCRIPTION:
Electrical storm (ES) is a life-threatening syndrome defined by the recurrence of ventricular arrythmias) and commonly occurs in implantable cardioverter defibrillator (ICD) recipients with an incidence ranging from 10 to 58% for secondary prevention. ES is also represented by a wide spectrum of clinical situations ranging from recurrent monomorphic VT reduced by anti-tachycardia pacing (ATP) in relatively stable patients to recurrent VF in hemodynamically unstable patients. Furthermore, ES can occur in the setting of acute reversible factors and/or underlying advanced structural heart disease. This wide clinical spectrum leads to major implications in ES management. Although several studies have focused on the predictors of ES and associated mortality, especially in the setting of VT ablation, only limited data assessing predictors of mortality following ES, are available. Thus, the purpose of this study was to assess the incidence and predictors of long term mortality following hospitalization in the intensive care unit for ES, in a large retrospective multicentric study.

ELIGIBILITY:
Inclusion Criteria:

All ventricular arrythmias admitted in ICU -

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted in ICU between january 2015 and june 2022
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Mortality | at 5 years

SECONDARY OUTCOMES:
Hospital duration | 0 to 30 day follow up

IPD SHARING:
Plan to Share IPD: No